CLINICAL TRIAL: NCT04905329
Title: Defendor Special: A Multicenter Prospective Observational Post-registration Study of Combined Chemotherapy With Empegfilrastim Support to Evaluate Safety and Efficacy in Patients With High and "Gray Zone" Risk Reccurrence Breast Cancer, Gastointestinal Cancers and Gynecological Malignancies
Brief Title: A Multicenter Prospective Post-registration Study of Empegfilgrastim to Evaluate Safety and Efficacy in Special Cancer Populations
Acronym: Def_Special
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Moscow Clinical Scientific Center (Other)
Responsible Party: Principal Investigator, Zhukova Lyudmila, Deputy Director of the Loginov Moscow Clinical Scientific Center, MD, PhD, Professor, Moscow Clinical Scientific Center
Other Study IDs: DS_v01
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumor; High-Risk Cancer; Breast Cancer; Gastrointestinal Cancer; Gynecological Malignancies; Myelosuppression
MeSH Terms: conditions — Breast Neoplasms; Gastrointestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with high and "gray zone" risk reccurrence early breast cancer
  Interventions: Drug: Empegfilgrastim
- Patients with gastointestinal cancers
  Interventions: Drug: Empegfilgrastim
- Patients with gynecological malignancies
  Interventions: Drug: Empegfilgrastim

INTERVENTIONS:
Drug: Empegfilgrastim — Extimia®

SUMMARY:
This study was designed to evaluate the efficacy and safety of Extimia® (INN - empegfilgrastim) in reducing the frequency, duration of neutropenia, the incidence of febrile neutropenia and infections caused by febrile neutropenia in patients with High and "Gray Zone" Risk Reccurrence Breast Cancer, Gastointestinal Cancers and Gynecological Malignancies

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Histologically verified diagnosis;
3. Age between 18 and 80 years; If the patient had previously received chemotherapy for these indications, then it should be completed at least 30 days before the first administration of the study drug;
4. ECOG performance 0-2;
5. Haematology:

   * ANC ≥ 1,5 х 10(9) /L;
   * Platelets ≥ 100 х 10(9) /L;
   * Hemoglobin ≥ 90 g/L;
6. Biochemistry:

   * Creatinine ≤ 1,5 ULN;
   * Total bilirubin ≤ 1,5 ULN;
   * AST/ALT ≤ 2,5 ULN;
   * Alkaline phosphatase ≤ 5 ULN;

8. Life expectancy of at least 6 months from the date of the first drug administration in the study; 9. Ability of the patient to comply with the Protocol requirements.

Exclusion Criteria:

1. Documented hypersensitivity to empegfilgrastim, filgrastim, pegfilgrastim, and / or their constituent excipients: pegylated drugs, protein recombinant drugs;
2. Systemic use of antibiotics less than 72 hours before the first drug administration in the study;
3. Concurrent or less than 30 days before the start of the study, radiation therapy (with the exception of point radiation therapy for bone metastases); study;
4. Concurrent participation in clinical trials, participation in clinical trials within the previous 30 days, previous participation in this study;
5. Surgical treatment less than 21 days (3 weeks) prior to study enrollment; taking any experimental medications less than 30 days before enrollment in this study;
6. History of bone marrow or hematopoietic stem cell transplantation;
7. Presence of acute or active chronic infections;
8. Other diseases (with the exception of the main one) that could affect the assessment of the severity of the symptoms of the underlying disease: that may mask, enhance, change the symptoms of the underlying disease or cause clinical manifestations and changes in the data of laboratory and instrumental research methods;
9. Inability to administer the drug by intravenous infusion or subcutaneous injection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with high and "gray zone" risk reccurrence breast cancer, gastointestinal cancers and gynecological malignancies who are prescribed myelosuppressive therapy with empegfilgrastim supportive therapy to support planned RDI, reduce the frequency, duration of neutropenia, the incidence of febrile neutropenia (FN) and infections manifested by FN, as part of routine clinical practice according to the approved indications of the appropriate drugs.
Sampling Method: Probability Sample
Enrollment: 285 (Estimated)
Dates: Start 2020-04-28 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Relative dose-intensity (RDI) of the myelosupressive therapy course | 12 months

SECONDARY OUTCOMES:
RDI of 6 x TC, 6 x TCHP, ddAC x4 -> 4 x paclitaxel , dd4AC -> 4 x paclitaxel + 12 x carboplatin) regimens performed in relation to (neo) adjuvant therapy of breast cancer | 18 months
RDI of FOLFOX-, FOLFOXIRI-based regimens performed in relation to (neo) adjuvant therapy of colorectal cancer | 18 months
RDI of FOLFOX-, FOLFOXIRI-based regimens performed in relation to patients with potentially resectable liver metastases of colorectal cancer | 18 months
RDI of DCF-, FOLFORINOX-based regimens performed in relation to therapy of pancreatic cancer | 18 months
RDI of DCF-, FOLFORINOX-, FLOT-, FOLFOX-based regimens performed in relation to therapy of gastric and esophageal cancers | 18 months
RDI of chemotherapy courses performed in patients with cervical cancer and sarcoma of the uterus after irradiation of the pelvic organs | 18 months
The complete pathological responses (pCR) rate in the primary tumors for patients diagnosed with HER2 + and triple negative early breast cancer requiring neoadjuvant treatment | 18 months
The complete pathological responses (pCR) rate in the malignant lymph nodes for patients diagnosed with HER2 + and triple negative early breast cancer requiring neoadjuvant treatment | 18 months
The incidence of febrile neutropenia with empegfilgrastim supportive therapy compared with historical control | 18 months
The incidence of neutropenia leading to a dose reduction of cytostatic drugs and / or an increase of the interval between cycles when using empegfilgrastim supportive therapy compared with historical controls | 18 months
Completed cases number of (neo) adjuvant therapy | 18 months
The incidence of severe infections (grade 3-4) | 18 months
Frequency of antibiotic prescription | 18 months
Frequency of study withdrawal due to adverse events | 18 months
RCB rate in patients with breast cancer | 18 months
Any grade adverse events frequency | 18 months
Serious adverse events frequency | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Inna Ganshina, MD, PhD, Principal Investigator — FSBI NMITs oncology named after N.N. Blokhin, the Ministry of Health of Russia; Lyudmila Zhukova, MD, PhD, professor, Study Chair — Moscow Clinical Scientific Center named after AS Loginov; Alexey Tryakin, MD, PhD, professor, Principal Investigator — FSBI NMITs oncology named after N.N. Blokhin, the Ministry of Health of Russia; Mikhail Fedyanin, MD, PhD, professor, Principal Investigator — FSBI NMITs oncology named after N.N. Blokhin, the Ministry of Health of Russia; Svetlana Khokhlova, MD, PhD, Principal Investigator — FSBI "National medical research center for obstetrics, gynecology and perinatology named after academician VI Kulakov" Ministry of healthcare of the Russian Federation
Locations (3):
- Russia (3):
  - Moscow Clinical Scientific Center named after AS Loginov, Moscow, Not Required
  - FSBI NMITs oncology named after N.N. Blokhin, the Ministry of Health of Russia, Moscow, Not Required
  - FSBI "National medical research center for obstetrics, gynecology and perinatology named after academician VI Kulakov" Ministry of healthcare of the Russian Federation, Moscow

IPD SHARING:
Plan to Share IPD: No